CLINICAL TRIAL: NCT00090532
Title: A Phase 1/2, Randomized, Masked, Single and Multiple-Dose, Sequential Dose-Escalation Study of the Safety an Efficacy of AG-013958 in Subjects With Subfoveal Choroidal Neovascularization Associated With Age-related Macular Degeneration
Brief Title: A Study Of The Safety And Efficacy Of AG-013,958 In Subjects With Subfoveal Choroidal Neovascularization Associated With Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to a lack of efficacy.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4321001
Record Dates: First submitted 2004-08-26; First posted 2004-08-31 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

INTERVENTIONS:
Drug: AG-013,958

SUMMARY:
AG-013,958 is being studied to treat patients with Age-Related Macular Degeneration. A total of 144 subjects may be enrolled in the trial. Subjects will be male or female at least 55 years of age with "wet" age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects >=55 years of age
* Subfoveal choroidal neovascularization complicating age-related macular degeneration
* Subjects who are informed of, and willing and able to comply with, the investigational nature of the study and are able to provide written informed consent in accordance with institutional and regulatory guidelines

Exclusion Criteria:

* Other serious ocular diseases or conditions, including diabetic retinopathy and glaucoma, that are likely to compromise visual acuity within 1 year

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155
Dates: Start 2004-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the ocular and systemic safety of the study drug

SECONDARY OUTCOMES:
To evaluate the visual acuity change after study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (30):
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Oro Valley, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Tuscon, Arizona
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Chevy Chase, Maryland
  - Pfizer Investigational Site, Hagerstown, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Livonia, Michigan
  - Pfizer Investigational Site, Rochester, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Saint Clair Shores, Michigan
  - Pfizer Investigational Site, Ypsilanti, Michigan
  - Pfizer Investigational Site, Slingerlands, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Lakewood, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Chambersburg, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Fairfax, Virginia
- Australia (2):
  - Pfizer Investigational Site, Sydney, New South Wales
  - Pfizer Investigational Site, East Melbourne, Victoria
- Netherlands (4):
  - Pfizer Investigational Site, Nijmegen, Gelderland
  - Pfizer Investigational Site, Amsterdam, North Holland
  - Pfizer Investigational Site, Groningen, Provincie Groningen
  - Pfizer Investigational Site, Rotterdam, South Holland
- United Kingdom (3):
  - Pfizer Investigational Site, Aberdeen, Scotland
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4321001&StudyName=A+Study+Of+The+Safety+And+Efficacy+Of+AG%2D013%2C958+In+Subjects+With+Subfoveal+Choroidal+Neovascularization+Associated+With+Age%2DRelated+Macular+Degeneration++